CLINICAL TRIAL: NCT02230358
Title: Cardiac Output and Cerebral Blood-flow During Carotid Endarterectomy in Regional vs. General Anesthesia. A Prospective Randomized Controlled Single Center Study
Brief Title: Cardiac Output and Duplex Sonography in Carotid Endarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Priv.Doz. Dr. Corinna Velik-Salchner, Priv.-Doz. Dr., Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CODUCE
Record Dates: First submitted 2014-07-31; First posted 2014-09-03 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Carotid Stenosis
Keywords: carotid endarterectomy; cardiac output; trans-cranial Doppler; CEA; regional anesthesia; general anesthesia
MeSH Terms: conditions — Carotid Stenosis | interventions — Anesthesia, Conduction; Anesthesia, General; Ultrasonography, Doppler, Transcranial; Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regional anesthesia (RA) (Other): Regional anesthesia (RA) for a carotid endarterectomy Interventions: Regional anesthesia (RA), blood gas analysis, 'Transcranieller Doppler' (Transcranial Doppler ultrasonography), invasive arterial blood pressure measurement, arterial blood gas measurement, neurological control, Near-infrared spectroscopy (NIRS) monitoring, oxygen supply (not invasive 'Vigileo')
  Interventions: Procedure: Regional anesthesia; Device: Transcranial Doppler ultrasonography; Procedure: blood gas analysis; Procedure: invasive arterial blood pressure measurement; Procedure: arterial blood gas measurement; Behavioral: Neurological Control; Behavioral: NIRS monitoring; Device: oxygen supply (not invasive 'Vigileo')
- General anesthesia (GA) (Other): General anesthesia (GA) for a carotid endarterectomy Interventions: General anesthesia, blood gas analysis, 'Transcranieller Doppler' (Transcranial Doppler ultrasonography), invasive arterial blood pressure measurement, arterial blood gas measurement, neurological control, NIRS monitoring, oxygen supply (not invasive 'Vigileo')
  Interventions: Procedure: General anesthesia; Device: Transcranial Doppler ultrasonography; Procedure: blood gas analysis; Procedure: invasive arterial blood pressure measurement; Procedure: arterial blood gas measurement; Behavioral: Neurological Control; Behavioral: NIRS monitoring; Device: oxygen supply (not invasive 'Vigileo')

INTERVENTIONS:
Procedure: Regional anesthesia — Regional anesthesia
  Arms: Regional anesthesia (RA)
Procedure: General anesthesia — General anesthesia
  Arms: General anesthesia (GA)
Device: Transcranial Doppler ultrasonography — 6x for 4 hours
Procedure: blood gas analysis — 6 x 3 ml blood withdrawal (18 ml) within 4 hours
Procedure: invasive arterial blood pressure measurement — before operation, 8 hours, as done in clinical routine
Procedure: arterial blood gas measurement — perioperative, 4-6 times within 8 hours, as done in clinical routine
Behavioral: Neurological Control — perioperative, 2-3 days, as done in clinical routine
Behavioral: NIRS monitoring — perioperative, for 5 hours, as done in clinical routine
Device: oxygen supply (not invasive 'Vigileo') — perioperative for 5 hours, as done in clinical routine

SUMMARY:
The aim of this study is to investigate the differences between the cardiac output and the cerebral blood-flow between a regional anesthesia (RA) and a general anesthesia (GA) in a randomized, controlled, single center study at the Medical University Innsbruck, Department of Anesthesia and Intensive Care Medicine.

DETAILED DESCRIPTION:
The investigators will investigate the differences between the cardiac output and the cerebral blood-flow between a regional anesthesia (RA) and a general anesthesia (GA) in a randomized, controlled, single center study at the Medical University Innsbruck, Department of Anesthesia and Intensive Care Medicine.

For this purpose patients with the need of a carotid endarterectomy (CEA) will be included and randomized either to the regional anesthesia (RA) or the general anesthesia (GA) group until a patient number of 45 in each group is achieved.

The cardiac output and cerebral blood-flow via trans-cranial Doppler (TCD) will be measured at 6 time points:

* T0 Baseline (after insertion of an arterial line)
* T1 After induction of anesthesia, but before surgical start
* T2 Two minutes after clamping the carotid artery
* T3 Two minutes after shunt insertation of the carotid artery
* T4 After reperfusion
* T5 After completion of the skin suture

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Elective carotid endarterectomy
3. Signed informed consent

Exclusion Criteria:

1. Age under 18 years
2. Missing signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Influence of anesthetic technique on cardiac output during carotid endarterectomy. | Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Number of participants: 90 patients
  Unit of measure: Cardiac index (l/m2)
  Cardiac output will be measured and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture

SECONDARY OUTCOMES:
Influence of anesthetic technique on trans-cranial doppler flow during carotid endarterectomy. | Change of cardiac output from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Cerebral blood flow will be measured via trans-cranial Doppler (TCD) and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture

OTHER OUTCOMES:
Influence of anesthetic technique on near infrared spectroscopy during carotid endarterectomy. | Change of cardiac output from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Number of participants: 90 patients
  Unit of measure: blood flow, volume and absolute tissue saturation
  Near infrared spectroscopy will be measured and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture
Influence of anesthetic technique on blood pressure during carotid endarterectomy. | Change of blood pressure, from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Number of participants: 90 patients
  Unit of measure: blood pressure in mmHg
  Blood pressure will be measured and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture
Percentage of participants with death. | Up to 6 months
Number of participants with transient ischemic attack and neck hematoma requiring surgical revision. | Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Percentage of participants with myocardial infarction. | Up to 6 months
Percentage of participants with stroke. | Up to 6 months
Influence of anesthetic technique on heart rate during carotid endarterectomy | Change of heart rate, from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Change of heart rate, from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Number of participants: 90 patients
  Unit of measure: beats per minute (bpm)
  Heart rate will be measured and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture
Influence of anesthetic technique on blood gas analysis during carotid endarterectomy | Change of oxygen saturation in blood, from Baseline to induction of anesthesia and up to 1 hour after admission to the intermediate care unit
  Number of participants: 90 patients
  Unit of measure: arterial oxygen tension (PaO2)
  Blood pressure will be measured and compared at the following time points:
  * T0 Baseline (after insertion of an arterial line)
  * T1 After induction of anesthesia, but before surgical start
  * T2 Two minutes after clamping the carotid artery
  * T3 Two minutes after shunt insertation of the carotid artery
  * T4 After reperfusion
  * T5 After completion of the skin suture

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Velik-Salchner, PrivDoz.Dr., Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria